CLINICAL TRIAL: NCT03163238
Title: The Effect of Dexmedetomidine on the Inflammatory Response in Children Under Congenital Heart Disease Repair With Cardiopulmonary Bypass: A Randomized Controlled Clinical Trial
Brief Title: Dexmedetomidine and the Inflammatory Response in Pediatric Cardiac Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Profossor of Anesthesiology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB000087632
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Cardiac Surgical Procedures
Keywords: Dexmedetomidine; Congenital Heart Disease; Cardiopulmonary Bypass; Interleukin
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Active Comparator): One syringe contain dexmedetomidine 0.5 mcg/kg diluted with normal saline in Dexmedetomidine group. Second syringe (50 ml) will contain normal saline (0.9%) in addition to Dexmedetomidine in addition to normal saline in Dexmedetomidine group. Concentration of Dexmedetomidine will be diluted according to the body weight so that we will fix the rate of infusion (1 ml/kg) to achieve a concentration of 0.5 mcg/kg/h in Dexmedetomidine group.
  Interventions: Drug: Dexmedetomidine
- Group S (Placebo Comparator): One syringe contain normal saline in 5 ml in Saline group. Second syringe (50 ml) will contain normal saline (0.9%) alone in rate of infusion (1 ml/kg) in Saline group
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.5 mcg/kg diluted with normal saline in Dexmedetomidine group. Second syringe (50 ml) will contain normal saline (0.9%) in addition to Dexmedetomidine in addition to normal saline in Dexmedetomidine group. Concentration of Dexmedetomidine will be diluted according to the body weight so that we will fix the rate of infusion (1 ml/kg) to achieve a concentration of 0.5 mcg/kg/h in Dexmedetomidine group.
  Other Names: Precedex
  Arms: Group D
Drug: Normal saline — One syringe contain normal saline in 5 ml in Saline group. Second syringe (50 ml) will contain normal saline (0.9%) alone in rate of infusion (1 ml/kg) in Saline group
  Other Names: Saline 0.9
  Arms: Group S

SUMMARY:
Cardiopulmonary bypass-assisted surgery initiates a systemic inflammatory response induced by extrinsic (e.g. anesthesia, contact activation within the extracorporeal circuit, endotoxemia) and intrinsic (e.g. tissue damage, endothelial cell activation, ischemia-reperfusion injury of myocardium) factors. This may either be mild or lead to a more severe clinical condition. Inflammation after pediatric open heart surgery is a parameter affecting also duration of mechanical ventilatory support. Dexmedetomidine use was associated with a reduced increase in plasma IL-1, IL-6, TNF-a, and INF-g levels

DETAILED DESCRIPTION:
Dexmedetomidine will be used during Cardiopulmonary bypass-assisted surgery for pediatric cardiac surgery

ELIGIBILITY:
Inclusion Elective repair of congenital heart disease with cardiopulmonary bypass Exclusion Reintervention surgery requirement for blood products from the start of CPB, preoperative intake of corticosteroids, deep hypothermia, those with preoperative low cardiac output, those with non-palpable peripheral pulses before surgery (e.g., accompanying coarctation of the aorta) or ischemic time during cardiopulmonary bypass more than 90 minutes

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Infilamatory response | Within the first 24 hours
  Interleukin 6 and 10

SECONDARY OUTCOMES:
Sedation score | Within the first 24 hours
  Special scale
Length of mechanical ventilaton | Within 7 days
  Length of mechanical ventilaton In days
Length of ICU stay | Within 7 days
  Length of ICU stay In days
Length of hospital stay. | Within 7 days
  Length of hospital stay days

CONTACTS AND LOCATIONS:
Overall Officials: Sayed K Abd-Elshafy, MD, Principal Investigator — Associate profossor of anesthesiology
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided